CLINICAL TRIAL: NCT07241247
Title: Clinical Study Evaluating the Role of Vitamin D Supplement in Patients With Colorectal Cancer Receiving Chemotherapy
Brief Title: Evaluation the of Role of Vitamin D Supplement on Tumor Response, Inflammation and Apoptosis in Patients With Stage II or III Colorectal Cancer Receiving Chemotherapy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Menna Allah Ayman Aboelenean, Clinical pharmacist, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2024ONCO15
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Vitamin D on Tumor Response and Inflammatory Markers; Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): (Vitamin D group; n=22) which will receive the same chemotherapy regimen plus Vitamin D for 6 months.
  Interventions: Drug: Vitamin D
- Control group (No Intervention): (Control group; n=22) which will receive FOLFOX (leucovorin, fluorouracil, and oxaliplatin) or XELOX (capecitabine and oxaliplatin).

INTERVENTIONS:
Drug: Vitamin D — Vitamin D supplement has effect on tumor response, inflammation and apoptosis
  Arms: Vitamin D group

SUMMARY:
The aim of this work is to assess the of role of Vitamin D supplement on tumor response, inflammation and apoptosis in patients with stage II or III colorectal cancer receiving chemotherapy using BAX protein and Tumor necrosis factor - alpha (TNF- α) both are measured at baseline and after 6 months.

DETAILED DESCRIPTION:
This randomized, controlled parallel study will be conducted on 44 patients with Stage II or III colorectal cancer. Patients will be recruited from Clinical Oncology

Department, Menoufia university Hospital, Menoufia, Egypt. The patients will be randomized using sealed envelope method into the following two groups:

Group I (Control group; n=22) which will receive FOLFOX (leucovorin, fluorouracil, and oxaliplatin) or XELOX (capecitabine and oxaliplatin).

Group II: (Vitamin D group; n=22) which will receive the same chemotherapy regimen plus Vitamin D for 6 months.

Markers to be measured:

* BAX protein as a marker for apoptosis will be measured at baseline and after 6 months.
* Tumor necrosis factor - alpha (TNF- α) as a marker of inflammation will be measured at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically and radiologically confirmed diagnosis of stage II or III colorectal cancer.
* Performance status 0-1 according to the Eastern Cooperative Oncology Group (ECOG).
* Patients who received FOLFOX or XELOX as first line chemotherapy.
* Both genders.
* Age ≥18.
* Patients with adequate hematologic parameters (white blood cell count ≥3000/mm3, granulocytes ≥1500/mm3, platelets ≥100,000/mm3, hemoglobin ≥ 8 gm/l).
* Patients with normal renal functions.
* Patients with normal hepatic functions.
* Patients with sufficient 25(OH) Vitamin D level (30-100 ng/mL).

Exclusion Criteria:

* Patients with metastatic colorectal cancer (CRC).
* Patients with parathyroid disorders.
* Patients who are taking vitamin D-containing supplements (>800 IU/day) unless they discontinued vitamin D supplementation at least 2 months prior to enrollment.
* Patients had a history of hypercalcemia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
The change in the serum concentrations of the measured biological markers | 6 months
  * BAX protein as a marker for apoptosis
  * Tumor necrosis factor - alpha (TNF- α) as a marker of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Menofia university, Cairo, Egypt